CLINICAL TRIAL: NCT07025395
Title: Development and Implementation of a Core Training Protocol: Effects on Muscle Activation, Hypertrophy, Balance, and Quality of Life in Recreationally Active Adults
Brief Title: "CORE Training for Musculoskeletal Health: A Study on Adaptive Exercise Protocols"
Acronym: RCT-EMG-US-QoL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ioannis Tsartsapakis (Other)
Responsible Party: Sponsor-Investigator, Ioannis Tsartsapakis, Laboratory Teaching Staff - Laboratory of Neuromechanics. Department of Physical Education and Sport Science at Serres, Aristotle University of Thessaloniki, Aristotle University Of Thessaloniki
Organization: Aristotle University Of Thessaloniki (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AUTH-CORE-STUDY
Record Dates: First submitted 2025-06-10; First posted 2025-06-17 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Core Muscle Weakness; Postural Control Deficit; Trunk Stability Impairment; Functional Performance Limitation
Keywords: Core Training; Neuromuscular Adaptations; Muscle Hypertrophy; Electromyography; Ultrasound Imaging; Functional Performance; Life Satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: This study employs a parallel-group design with randomized allocation. Participants are divided into an experimental group undergoing an eight-week core training protocol and a control group following a standardized core-related routine. The interventional group receives structured progressive stability, strength, and power-focused exercises, while the control group engages in general core activation without targeted neuromuscular training. Pre- and post-intervention assessments evaluate neuromuscular function, balance, biomechanical efficiency, and life satisfaction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group - Progressive Core Training Protocol (Experimental): Participants in this arm will follow an eight-week structured core training protocol designed to enhance neuromuscular adaptations, core muscle hypertrophy, and biomechanical performance. The program incorporates progressive core stability, core strength, and high-intensity core power exercises, ensuring gradual intensity scaling and optimized movement efficiency. Training sessions include warm-up, eight structured triads of core exercises, and a cool-down phase. Assessments will track electromyographic activity, ultrasound muscle imaging, balance performance, and kinetic chain optimization.
  Interventions: Behavioral: - Core Training Protocol
- Control Group - Standardized Core Routine (Active Comparator): Participants in this arm will engage in a standardized core exercise routine performed twice per week. The intervention will not include progressive intensity or specialized neuromuscular activation techniques. Control group participants will perform basic abs and back exercises to maintain general core function without targeted adaptations. The purpose of this arm is to serve as a baseline comparison for neuromuscular, biomechanical, and psychological assessments between groups.
  Interventions: Behavioral: Control Group Core Routine

INTERVENTIONS:
Behavioral: - Core Training Protocol — This structured training intervention incorporates progressive core exercises designed to enhance neuromuscular activation, balance, and muscle hypertrophy. Participants perform eight exercise triads per session, progressing from core stability drills to high-intensity power movements over eight weeks.
  Arms: Experimental Group - Progressive Core Training Protocol
Behavioral: Control Group Core Routine — Control group participants engage in general core activation exercises twice per week, without progressive intensity or specialized neuromuscular adaptation.
  Arms: Control Group - Standardized Core Routine

SUMMARY:
This study aims to evaluate the effects of an adaptive core training protocol that integrates core stability, core strength, and high-intensity core power exercises on muscle activation, hypertrophy, balance, and quality of life. Forty recreationally active adults with a minimum of two years of consistent training experience will participate. The structured intervention will span multiple weeks and utilize electromyography (EMG), ultrasound imaging, and validated questionnaires to assess neuromuscular and functional adaptations.

DETAILED DESCRIPTION:
Extended Detailed Description - Study Rationale and Objectives Core stability is a foundational component of human movement, contributing to postural control, balance, and force transmission. The deep and superficial muscle systems of the trunk function synergistically to enhance spinal alignment, movement efficiency, and musculoskeletal integrity.

In modern health science, core training has evolved into a key preventative strategy that supports spinal resilience and reduces functional limitations associated with sedentary lifestyles. Contemporary protocols often integrate trunk bracing, diaphragmatic engagement, and multi-planar control for comprehensive development.

This randomized, controlled trial evaluates the effects of an eight-week progressive core training program in recreationally active adults. The protocol combines components of neuromuscular control, strength development, and high-intensity power work, and aims to assess outcomes related to muscle activation, balance, segmental coordination, and perceived well-being.

Study Design & Participants Participants will be randomly assigned to an experimental group (receiving the full protocol) or a control group (minimal activity). All procedures will take place at the Neuromechanics Laboratory of the Aristotle University of Thessaloniki (Serres Campus). Forty adults between 25-35 years old who meet physical activity and health-related eligibility criteria will complete baseline and post-intervention assessments. Written informed consent will be obtained prior to randomization.

Core Training Structure The program consists of a warm-up (~6 min), a main core-focused session (~30-32 min), and a cool-down (~5 min). Training follows a triad structure in which each set includes one stability, one strength, and one power-based core exercise. Work intervals are set to 45 seconds, with progressive recovery. All sessions are designed to follow a logical kinetic chain progression: from motor control to peak force expression.

Measurements & Instrumentation Pre- and post-testing includes validated assessments of ground reaction force, muscle activation, ultrasound-measured hypertrophy, video-based kinematic analysis, body measurements, and psychometric indices of well-being. Instrumentation includes force platforms, surface EMG, ultrasound imaging systems, motion capture tools, and standardized questionnaires.

Anticipated Outcomes The intervention is expected to improve neuromuscular efficiency, postural control, force production, core muscle thickness, and overall movement confidence. Enhanced trunk function may contribute to greater kinetic chain integration and better quality of life.

Broader Impact and Applicability Due to its equipment-light structure and progressive difficulty, this training protocol is well-suited for application in clinical rehabilitation, fitness centers, or at-home settings under professional supervision. The triad design offers educational value for exercise professionals seeking to integrate functional core sequencing into their practice.

This trial contributes to ongoing research on motor control strategies, force adaptation, sensorimotor integration, and holistic well-being. Insights gained may inform interventions in athletic populations, workplace health promotion, and functional aging.

ELIGIBILITY:
Inclusion Criteria:

* Aged 25-35 years
* Physically active (≥3 sessions/week, ≥1 hour per session) for ≥2 years
* No known musculoskeletal, cardiovascular, or neurological disorders
* No engagement in structured core training programs
* Available to attend all evaluation appointments
* Able and willing to commit to the 8-week intervention program

Exclusion Criteria:

* Medical conditions that limit full-body or trunk movement
* Cardiovascular/metabolic conditions contraindicating high-intensity exercise
* Current participation in Pilates, CrossFit, or other core-specific protocols
* Recent musculoskeletal injury affecting training eligibility

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Electromyographic (EMG) Muscle Activation During Medicine Ball Overhead Slam | Baseline (Week 0) and Post-Intervention (Week 8)
  Surface EMG recordings will assess neuromuscular activation in the rectus abdominis (RA), external oblique (EO), and iliocostalis lumborum (IL) muscles. Measurements will be conducted pre- and post-intervention using Biopac Systems Inc. electrodes and TEL100 M transmitter, with signals filtered between 10-500 Hz. Data will be analyzed via Acknowledge software to determine training-induced improvements in core muscle activity patterns.

SECONDARY OUTCOMES:
Ultrasound-Based Core Muscle Hypertrophy Assessment | Baseline (Week 0) and Post-Intervention (Week 8)
  B-mode ultrasound imaging (Aloka ProSound SSD 3500 SV) will evaluate changes in muscle thickness of the transverse abdominis (TrA), internal oblique (IO), and lumbar multifidus (LM) at rest. Pre- and post-intervention measurements will quantify hypertrophic adaptations induced by structured core training."
Balance & Postural Stability Evaluation (Force Plate Analysis) | Baseline (Week 0) and Post-Intervention (Week 8)
  Static and dynamic balance assessments will be conducted using a Kistler 3D dynamometer, with center-of-pressure displacement analyzed pre- and post-intervention. Improvements in balance metrics are expected to reflect enhanced neuromuscular control and stability.
Psychometric Evaluation of Life Satisfaction (Satisfaction With Life Scale - SWLS) | Baseline (Week 0) and Post-Intervention (Week 8)
  The Satisfaction With Life Scale (SWLS) will be used to assess subjective well-being before and after the intervention. The scale consists of 5 items scored on a 7-point Likert scale. Total scores range from 5 to 35, with higher scores indicating greater life satisfaction.

OTHER OUTCOMES:
Kinematic Angular Velocity Analysis (Motion Capture) | Baseline (Week 0) and Post-Intervention (Week 8)
  High-definition motion tracking will quantify angular velocity changes in shoulder, hip, and knee joints during medicine ball overhead slams. Assessments will be performed using a PTZOptics Move 4K camera and Kinovea biomechanics software.
Psychometric Evaluation of Life Satisfaction (SWLS) | Baseline (Week 0) and Post-Intervention (Week 8)
  The Satisfaction With Life Scale (SWLS) will be administered pre- and post-intervention to assess subjective well-being and psychological benefits associated with neuromuscular training adaptations."

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Tsartsapakis, Ph.D., Principal Investigator — Aristotle University of Thessaloniki, Greece
Locations (1):
- Aristotle University of Thessaloniki, Serres Campus - Neuromechanics Laboratory, Serres, Central Makedonia, Greece

IPD SHARING:
Plan to Share IPD: Undecided
Currently, there are no plans to share individual participant data (IPD). However, anonymized datasets may be made available upon institutional approval for future research focusing on neuromuscular adaptations, biomechanics, and core training effects.

REFERENCES:
- See also: Department of Physical Education and Sport Science at Serres AUTH — https://phed-sr.auth.gr/%CF%84%CE%BC%CE%AE%CE%BC%CE%B1-%CE%B5%CF%80%CE%B9%CF%83%CF%84%CE%AE%CE%BC%CE%B7%CF%82-%CF%86%CF%85%CF%83%CE%B9%CE%BA%CE%AE%CF%82-%CE%B1%CE%B3%CF%89%CE%B3%CE%AE%CF%82-%CE%B1%CE%B8%CE%BB%CE%B7%CF%84%CE%B9%CF%83%CE%BC%CE%BF%CF%8D-%CF%83%CE%B5%CF%81%CF%81%CF%8E%CE%BD-%CE%B1%CF%80%CE%B8
- Available data/document: Study Protocol: 28 May 2025 — https://youtu.be/ql8SD07abnI — Core Training Protocol by Ioannis Tsartsapakis Ph.D.